CLINICAL TRIAL: NCT06757452
Title: The Effect of Supplementation with Curcuminoids for the Improvement of Musculoskeletal Conditions in Sedentary Adults
Acronym: curcuminoids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lissette Ariza Corredor (Industry)
Collaborators: Universidad de Caldas (Other)
Responsible Party: Sponsor-Investigator, Lissette Ariza Corredor, R&D Manager, Inbiotech
Organization: Inbiotech (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CBCS-030
Record Dates: First submitted 2024-12-19; First posted 2025-01-03 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Sedentariness and Well-being
Keywords: curcuminoid; sedentarism; recovery; inflammation; antioxidants
MeSH Terms: conditions — Inflammation | interventions — Diarylheptanoids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Experimental unit who received Placebo were treated equaly as the supplemented group.
  The control group received a placebo capsule of 250 mg maltodextrin.
  Interventions: Other: Physical excercise
- Supplemented (Experimental): who received Cal LX. Cal LX is a food-grade dietary supplement based on turmeric, it has been designed to improve physical resistance during exercise, accelerate post-exercise recovery, and reduce the feeling of muscle soreness. Cal LX was determined as not cytotoxic or genotoxic. The supplement or placebo dosage was one (1) 250 mg capsule 45 minutes before exercising.
  Interventions: Dietary Supplement: Supplement with curcuminoids; Other: Physical excercise

INTERVENTIONS:
Dietary Supplement: Supplement with curcuminoids — Cal LX is a food-grade dietary supplement based on turmeric, it has been designed to improve physical resistance during exercise, accelerate post-exercise recovery, and reduce the feeling of muscle soreness. Cal LX was determined as not cytotoxic or genotoxic. The supplement or placebo dosage was one (1) 250 mg capsule 45 minutes before exercising.
  Other Names: Cal LX
  Arms: Supplemented
Other: Physical excercise — Participants performed 45 minutes of physical activity twice a week. The intervention program included a five-minute warm-up, composed of two series of joint mobility and three series of eight seconds of lower limbs stretching. Then, a routine of intermittent training composed of four six-minute rounds was directed. Each routine included running for 10 seconds and a pause between them. The first round had a 20 s pause, the second round 15 s, and the third and fourth rounds 10 s. Between the rounds was a two-minute passive pause. Finally, three series of twenty seconds of elongation of the lower extremities were required as colling down.

SUMMARY:
The aim of this study is to evaluate the effect of a supplementation with curcuminoids, called Cal LX, prior to physical exercise, on the improvement of musculoskeletal conditions in sedentary people, which would lead to more physical exercise regularly.

ELIGIBILITY:
Inclusion Criteria:

* To be over 25 years old
* To have not exercised systematically during the last 3 months, or do not do physical exercise daily for more than 25 minutes per day for a maximum of 3 days per week
* Sitting for at least 4 hours continuously
* Type 2 diabetes patients.

Exclusion Criteria:

* To have a history or diagnoses of cardiopulmonary, osteoarticular, type 1 diabetes or autoimmune disorders
* Pregnancy
* Smokers.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
RMSSD | Twice a week, prior and after the physical activity, during the three monts of intervention
  An indicator of parasympathetic activity by evaluating the root mean square of successive differences between normal heartbeats (RMSSD) determined in milliseconds, which is directly associated with short-term heart rate variability.

SECONDARY OUTCOMES:
Creatinine | Every 30 days, begining the first day physical activity, during the three monts of intervention.
  Creatinine is a waste product that comes from the digestion of protein in your food and the normal breakdown of muscle tissue. It is removed from the blood through your kidneys.
CK | Every 30 days, begining the first day physical activity, during the three monts of intervention.
  Creatine kinase is an enzyme that's responsible for healthy muscle function. When muscles break down, they release CK, elevating the protein levels in your blood.
LDH | Every 30 days, begining the first day physical activity, during the three monts of intervention.
  LDH is an enzyme found in many body tissues such as the heart, liver, kidney, skeletal muscle, brain, blood cells, and lungs. When body tissue is damaged, LDH is released into the blood.
Urea | Every 30 days, begining the first day physical activity, during the three monts of intervention.
  Urea and creatinine levels are used to evaluate kidney function.
SOD | Every 30 days, begining the first day physical activity, during the three monts of intervention.
  Superoxide dismutase (SOD) is an enzyme found in all living cells. An enzyme is a substance that speeds up certain chemical reactions in the body. Superoxide dismutase helps break down potentially harmful oxygen molecules in cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Caldas, Manizales, Caldas Department, Colombia

IPD SHARING:
Plan to Share IPD: No